CLINICAL TRIAL: NCT04866290
Title: Prospective Registry of Transarterial Chemoembolization of Metastatic Colorectal Cancer to the Liver With HepaSphere™ Microspheres Loaded With Irinotecan
Brief Title: HepaSphere™ Microspheres Prospective Registry
Acronym: mCRC
Status: Completed | Type: Observational
Sponsor: Merit Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CRC-P4-16-01
Record Dates: First submitted 2021-04-27; First posted 2021-04-29 (Actual); Results first posted 2022-10-12 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Colorectal Cancer; Liver metastases; Transarterial chemoembolization
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: HepaSphere Microspheres

SUMMARY:
HepaSphere™ Microspheres loaded with irinotecan received CE mark for the indication of use in embolization of metastatic colorectal cancer (mCRC) to the liver in 2015.

The purpose of this registry is to demonstrate the safety and efficacy of HepaSphere Microspheres loaded with irinotecan for the treatment of colorectal liver metastasis and add to the understanding of the use and value of this treatment in 'real life' usage conditions.

DETAILED DESCRIPTION:
This prospective, post-market study was designed to evaluate the median overall survival (MOS) of subjects with metastatic colorectal cancer (mCRC) to the liver treated with HepaSphere Microspheres loaded with the chemotherapeutic agent irinotecan. This treatment process is referred to as transarterial chemoembolization (TACE).

Subjects with confirmed colorectal cancer liver metastases that were ineligible for surgical hepatic tumor resection and that had not undergone prior TACE for this indication were considered for study participation. Patients that met eligibility criteria, wanted to participate in the study, and signed the informed consent form (ICF) made up the study subject population. All study subjects were in one cohort and were not blinded to treatment.

Per protocol, all subjects completed a baseline visit to collect medical history information, lab assessments, and have a baseline MRI. Following this baseline visit subjects were to have two TACE cycles (i.e., TACE Cycle 1, TACE Cycle 2), with TACE Cycle 2 occurring within 2-4 weeks following TACE Cycle 1. A TACE cycle is defined as one TACE procedure for subjects with unilobar disease or two TACE procedures for subjects with bilobar disease (i.e., one for each lobe of the liver). Following completion of TACE Cycle 1 and TACE Cycle 2, additional TACE cycles could be performed at the investigator's discretion for residual or new disease.

When subjects had completed two TACE cycles and were no longer indicated for further TACE cycles (at the investigator's discretion), they entered follow-up. The study ended and analysis began when all enrolled subjects had (1) completed two-year (24 months) follow-up from the date of TACE Cycle 1, (2) been deemed lost to follow up, or (3) died, whichever occurred first.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or radiologically confirmed colorectal cancer metastases to the liver
* Patient is able to have either CT or MRI imaging
* Hepatic tumor burden ≥50% of total tumor burden
* Hepatic tumor burden ≤50% of total liver volume
* Not suitable for treatment by resection or percutaneous ablation at time of TACE treatment
* Life expectancy ≥ 3 months
* WHO performance status ≤ 2

Exclusion Criteria:

* Previous treatment with any form of hepatic transarterial embolization
* Total bilirubin ≥ 3.0 mg/dL
* Any contraindication for irinotecan administration
* Partial or complete thrombosis of the main portal vein
* Cardiovascular or respiratory failure
* Any other condition deemed exclusionary by the Investigator

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with unresectable metastatic colorectal cancer with metastases to the liver.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2016-09-22 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katerina Malagari, MD, Principal Investigator — Evgenidio Hospital/ATTIKO Hospital
Locations (2):
- European Hospital Georges Pompidou, Paris, France
- Evgenidio Hospital/ATTIKO Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study enrollment began in September 2016 and ended in May 2019.
Groups:
- Patients With Metastatic Colorectal Cancer to the Liver: This was a non-randomized, single arm, prospective study that included all enrolled study participants that met the inclusion criteria, did not meet the exclusion criteria, and provided written informed consent.
Period: Enrolled and Completion of TACE Cycle 1
Arm/Group | Patients With Metastatic Colorectal Cancer to the Liver
Started | 105
Completed | 105
Not Completed | 0
Period: Completion of TACE Cycle 2
Arm/Group | Patients With Metastatic Colorectal Cancer to the Liver
Started | 105
Completed | 58
Not Completed | 47

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Metastatic Colorectal Cancer to the Liver
Number analyzed (Participants) | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 83
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Greece | 100
  France | 5
Baseline Disease Status: Tumor Location [Count of Participants; unit: Participants]
  Unilobar Liver Disease/Tumor Location | 65
  Bilobar Liver Disease/ Tumor Location | 40

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Median overall survival of subjects treated with HepaSphere Microspheres loaded with irinotecan. Analysis will be performed when all subjects enrolled have been followed for survival for two years (24 months), are considered lost to follow up, or have died, whichever comes first
Time Frame: 24 months
Population: All enrolled subjects received one or more TACE Cycles and therefore were included in the calculation of the primary endpoint, Median Overall Survival.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Patients With Metastatic Colorectal Cancer to the Liver
Number analyzed (Participants) | 105
months | 19 [14.0 to 23.0]

2. Secondary Outcome: Objective Response Rate (ORR)
Description: Determined by the Modified Response Evaluation Criteria In Solid Tumors Criteria (mRECIST) when all subjects enrolled have been followed for survival for 2 years (from date of 1st TACE), are considered lost to follow up, or have died, whichever comes first. Per mRECIST (target lesions assessed by MRI): Complete Response (CR), at least >=30% decrease in the sum of diameters of all viable target lesions, Partial Response (PR), at least a >=30% decrease in the sum of diameters of all viable target lesions, Stable Disease (SD), any cases that do not qualify for either partial response or progressive disease, Progressive Disease (PD), An increase of at least 20% in the sum of the diameters of or viable (enhancing) target lesions, taking as reference the smallest sum of the diameters of viable (enhancing) target lesions recorded since started. Overall Response (OR) = CR + PR. ORR is calculated as= (no. of patients with CR + the no. of patients with PR) / N. (N= No of participants analyzed)
Time Frame: 24 months
Population: Only subjects with complete imaging could be analyzed. Eighty three of the subjects had imaging and were evaluated using mRECIST criteria to calculate the objective response rate (ORR).
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Metastatic Colorectal Cancer to the Liver
Number analyzed (Participants) | 83
Participants
  Complete Response (CR) | 5
  Partial Response (PR) | 30

3. Secondary Outcome: Best Tumor Response
Description: Per the Modified Response Evaluation Criteria In Solid Tumors Criteria (mRECIST) for target lesions and assessed by MRI: Complete Response (CR), at least > =30% decrease in the sum of diameters of all viable ( enhancement in the arterial phase) target lesions, Partial Response (PR), at least a >=30% decrease in the sum of diameters of all viable (enhancement in the arterial phase) target lesions, Stable Disease (SD), any cases that do not qualify for either partial response or progressive disease, Progressive Disease (PD), An increase of at least 20% in the sum of the diameters of or viable (enhancing) target lesions, taking as reference the smallest sum of the diameters of viable (enhancing) target lesions recorded since started.
  Best Tumor Response (BTR) was assessed during the period of time between TACE Cycle 1 and the last post-TACE MRI or CT. BTR will be presented as the number of subjects within each response category and percentage of evaluated subjects.
Time Frame: 24 months
Population: Only subjects with complete imaging could be analyzed. Eighty three of the subjects had imaging and were evaluated using mRECIST criteria.
Measure: Count of Participants; unit: Participants
Groups:
- Patients With Metastatic Colorectal Cancer to the Liver: This was a non-randomized, single arm, prospective study that included all enrolled study participants that met the inclusion criteria, did not meet the exclusion criteria, and provided written informed consent.
  Best Tumor Response (BTR) was evaluated in 83 subjects using mRECIST criteria.
Arm/Group | Patients With Metastatic Colorectal Cancer to the Liver
Number analyzed (Participants) | 83
Participants
  Complete Response (CR) | 5
  Partial Response (PR) | 30
  Stable Disease (SD) | 25
  Progressive Disease (PD) | 23

4. Secondary Outcome: Liver Progression-free Survival
Description: Median liver progression-free survival will be calculated as the time (in months) between the first TACE procedure to the date on which progression of the subject's liver metastases was documented or the date of death (from any cause).
  Per the Modified Response Evaluation Criteria In Solid Tumors Criteria (mRECIST) for target lesions and assessed by MRI, Progressive Disease (PD) is defined as an increase of at least 20% in the sum of the diameters of or viable (enhancing) target lesions, taking as reference the smallest sum of the diameters of viable (enhancing) target lesions recorded since started.
Time Frame: 24 months
Population: Only 17 subjects had data available to calculate progression free survival (definition: a lack of tumor progression in the liver as determined by mRECIST criteria).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Patients With Metastatic Colorectal Cancer to the Liver
Number analyzed (Participants) | 17
months | 4.0 [3.00 to NA] — NA Explanation: The confidence interval cannot be calculated for the upper bounds of median survival because less than 50% of events (e.g. alive, death) have occurred from the low sample of 17 subjects. The upper limit of the survival curve has not reached 50% and thus, there is no estimate for the upper confidence limit on the median.

5. Secondary Outcome: Time to Progression
Description: Time to Progression (TTP) was defined as the length of time between TACE Cycle 1 and disease progression (as determined by MRI or CT imaging) of both hepatic and extrahepatic disease. The date of the first study TACE was time zero.
Time Frame: 24 months
Population: A total of 87 subjects had disease progression after one or more study TACE procedures, 66 with hepatic progression and 21 with extrahepatic progression.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Patients With Metastatic Colorectal Cancer to the Liver
Number analyzed (Participants) | 87
Months
  Hepatic Liver Disease: number analyzed (Participants) | 66
  Hepatic Liver Disease | 7.0 [6.0 to 9.0]
  Extra Hepatic Disease: number analyzed (Participants) | 21
  Extra Hepatic Disease | 6.0 [3.0 to 9.0]

ADVERSE EVENTS:
Time Frame: Treatment related adverse events (AEs) were collected throughout the duration of this study. Follow-up ranged from 30 to 1315 days.
Description: Only treatment related adverse events (AEs) were collected throughout the duration of this study. Treatment related AEs were defined as AEs that occurred on the day of or any day following a subject's first TACE procedure and determined to be treatment related by the investigator.
Arm/Group | Patients With Metastatic Colorectal Cancer to the Liver
All-Cause Mortality (participants affected / at risk) | 79/105
Serious Adverse Events (participants affected / at risk) | 1/105
Other Adverse Events (participants affected / at risk) | 97/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Metastatic Colorectal Cancer to the Liver (N=105)
Tumor rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Metastatic Colorectal Cancer to the Liver (N=105)
Abdominal pain upper (Gastrointestinal disorders) | 89 (180)
Nausea (Gastrointestinal disorders) | 28 (31)
Vomiting (Gastrointestinal disorders) | 19 (20)
Fatigue (General disorders) | 17 (18)
Pyrexia (General disorders) | 4 (5)
Abscess (Infections and infestations) | 1 (1)
Liver abscess (Infections and infestations) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Blood bilirubin increased (Investigations) | 12 (16)
Hepatic enzyme increased (Investigations) | 1 (1)
Transaminases increased (Investigations) | 10 (12)
White blood cell count increased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-04-21): https://cdn.clinicaltrials.gov/large-docs/90/NCT04866290/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-08): https://cdn.clinicaltrials.gov/large-docs/90/NCT04866290/SAP_001.pdf